CLINICAL TRIAL: NCT03821558
Title: Cardiovascular Rehabilitation in Coronary Artery Disease Patients: Influence of Different Types of Exercise Training on Selected Cardiovascular Parameters
Brief Title: Exercise Training in Individuals With Coronary Artery Disease
Acronym: ReKoBo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Borut Jug, Associate Professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKCLRehab0012019
Record Dates: First submitted 2019-01-06; First posted 2019-01-30 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Coronary Artery Disease; Myocardial Infarction
Keywords: exercise; interval training; continuous training; endothelial dysfunction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval training group (Active Comparator): Patients to be randomized to the 'interval training group' will have exercise training sessions 3 times per week for a period of 12 weeks. During training, they will undergo interval exercise series composed of high-intensity intervals (80-90% of peak exercise performance) and low-intensity intervals (60-70% of peak exercise performance).
  Interventions: Other: Exercise training
- Continuous training group (Active Comparator): Patients to be randomized to the 'continuous training group' will have exercise training sessions 3 times per week for a period of 12 weeks. During training, they will undergo moderate continuous exercise training at 75% of peak exercise performance.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Patients to be randomized to the 'interval training group' or 'continuous training group' will undergo exercise training sessions with different intensity levels.

SUMMARY:
In this controlled trial, patients referred to post-myocardial infarction cardiac rehabilitation will be randomized to either interval or continuous training.

DETAILED DESCRIPTION:
The trial would i) compare the acute effects of each exercise type on selected cardiovascular indicators; ii) compare the chronic effects of each exercise type on selected cardiovascular indicators; iii) provide information on the association between acute and chronic effects of each exercise type; iv) provide insight into possible mechanisms of effectiveness of each exercise type; v) identify the most safe and effective exercise type for patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* myocardium infarction 120 days prior to cardiac rehabilitation

Exclusion Criteria:

* contraindications for exercise training,
* uncontrolled dysrhythmias,
* uncontrolled heart failure (New York Heart Association (NYHA) stage IV),
* intellectual development disorder,
* pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Change of flow-mediated dilatation of the brachial artery, measured in % | 3 months

SECONDARY OUTCOMES:
Change of the arterial stiffness coefficient | 3 months
Change of maximal oxygen uptake during exercise, measured in ml/kg/min | 3 months
Change of the heart rate variability | 3 months
Change of the heart rate recovery | 3 months
Change in health-related quality of life using SF-36 questionnaire, measured in points | 3 months
  It is a self-administered questionnaire comprising 36 items measuring eight dimensions and two subscales (physical and mental)
Change in IL-6, IL-8, IL-10, TNF-alpha and NT-proBNP levels, measured in ng/l | 3 months
Change in osteopontin and D-dimer levels, measured in microg/l | 3 months
Change in selectin and hsCRP, measured in mg/l | 3 months
Change in hsTnI, CK MB, endocan, sST2, galectin-3, NGAL, CD40 ligand and BDNF, measured in ng/l | 3 months
Change in copeptin levels, measured in pmol/l | 3 months
Change in MR-proADM and MR-proANP, measured in nmol/l | 3 months
Change in homoarginine, ADMA and SDMA levels, measured in micromol/l | 3 months
Change in fibrinogen and Lp(a) levels, measured in mg/dl | 3 months
Change in insuline level, measure in microIU/ml | 3 months
Change in total cholesterol, LDL, HDL, triglycerides and glucose levels, measured in mmol/l | 3 months
Change in overall haemostatic potential | 3 months

OTHER OUTCOMES:
Change in the flow-mediated dilation during single exercise training session, measured in % | 3 months
Change in IL-6, IL-8, IL-10, TNF-alpha and NT-proBNP levels during single exercise training session, measured in ng/l | 3 months
Change in selectin and hsCRP during single exercise training session, measured in mg/l | 3 months
Change in hsTnI, CK MB, endocan, sST2, galectin-3, NGAL, CD40 ligand and BDNF levels during single exercise training session, measured in ng/l | 3 months
Change in copeptin levels during single exercise training session, measured in pmol/l | 3 months
Change in homoarginine, ADMA and SDMA levels during single exercise training session, measured in micromol/l | 3 months
Change in fibrinogen level during single exercise training session, measured in mg/dl | 3 months
Change in insuline levels during single exercise training session, measure in microIU/ml | 3 months
Change in osteopontin and D-dimer levels during single exercise training session, measured in microg/l | 3 months
Change in overall haemostatic potential during single exercise training session | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Borut Jug, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726
- [Background] Liou K, Ho S, Fildes J, Ooi SY. High Intensity Interval versus Moderate Intensity Continuous Training in Patients with Coronary Artery Disease: A Meta-analysis of Physiological and Clinical Parameters. Heart Lung Circ. 2016 Feb;25(2):166-74. doi: 10.1016/j.hlc.2015.06.828. Epub 2015 Jul 22. PMID 26375499
- [Background] Conraads VM, Pattyn N, De Maeyer C, Beckers PJ, Coeckelberghs E, Cornelissen VA, Denollet J, Frederix G, Goetschalckx K, Hoymans VY, Possemiers N, Schepers D, Shivalkar B, Voigt JU, Van Craenenbroeck EM, Vanhees L. Aerobic interval training and continuous training equally improve aerobic exercise capacity in patients with coronary artery disease: the SAINTEX-CAD study. Int J Cardiol. 2015 Jan 20;179:203-10. doi: 10.1016/j.ijcard.2014.10.155. Epub 2014 Oct 25. PMID 25464446
- [Background] Villelabeitia-Jaureguizar K, Vicente-Campos D, Senen AB, Jimenez VH, Garrido-Lestache MEB, Chicharro JL. Effects of high-intensity interval versus continuous exercise training on post-exercise heart rate recovery in coronary heart-disease patients. Int J Cardiol. 2017 Oct 1;244:17-23. doi: 10.1016/j.ijcard.2017.06.067. Epub 2017 Jun 17. PMID 28648356
- [Background] Currie KD, Rosen LM, Millar PJ, McKelvie RS, MacDonald MJ. Heart rate recovery and heart rate variability are unchanged in patients with coronary artery disease following 12 weeks of high-intensity interval and moderate-intensity endurance exercise training. Appl Physiol Nutr Metab. 2013 Jun;38(6):644-50. doi: 10.1139/apnm-2012-0354. Epub 2013 Jan 17. PMID 23724882
- [Background] Novakovic M, Prokselj K, Rajkovic U, Vizintin Cuderman T, Jansa Trontelj K, Fras Z, Jug B. Exercise training in adults with repaired tetralogy of Fallot: A randomized controlled pilot study of continuous versus interval training. Int J Cardiol. 2018 Mar 15;255:37-44. doi: 10.1016/j.ijcard.2017.12.105. Epub 2018 Jan 3. PMID 29338917